CLINICAL TRIAL: NCT06287931
Title: Probiotics for Gallstones in Post-bariatric Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Linglong Yingcheng Hospital (Network)
Responsible Party: Principal Investigator, Xuan Qiu, MD, Shandong Linglong Yingcheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: sdllycyy001
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery Candidate; Gallstone; Gallstone Attack; Gastrointestinal Quality of Life Index; Probiotics
Keywords: Bariatric Surgery Candidate; Gallstone; Probiotics
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ursodoxycholic acid group (Experimental): Ursodoxycholic acid, 250mg po tid x 6 months
  Interventions: Drug: Ursodoxycholic acid group
- Bifidobacterium group (Experimental): Bifidobacteria, 210 mg po tid x 6 months
  Interventions: Drug: Bifidobacterium group
- Bifidobacterium and ursodeoxycholic acid group (Experimental): Ursodoxycholic acid, 250mg po tid x 6 months Bifidobacteria, 210 mg po tid x 6 months
  Interventions: Drug: Ursodoxycholic acid group; Drug: Bifidobacterium group

INTERVENTIONS:
Drug: Ursodoxycholic acid group — Ursodoxycholic acid, 250mg po tid x 6 months
  Arms: Bifidobacterium and ursodeoxycholic acid group; Ursodoxycholic acid group
Drug: Bifidobacterium group — Bifidobacteria, 210 mg po tid x 6 months
  Arms: Bifidobacterium and ursodeoxycholic acid group; Bifidobacterium group

SUMMARY:
Obesity is an increasing epidemic worldwide and has a significant impact on human health and socioeconomics. Multiple studies have shown that bariatric surgery increases the risk of postoperative gallbladder stones. Contributing factors to gallstone formation include gallbladder motility and bile supersaturation due to rapid weight loss and cholesterol mobilization. At present, the prevention and treatment of gallbladder stones in obese patients after bariatric surgery are still controversial. In recent years, the study of ursodeoxycholic acid in preventing gallbladder stone formation after bariatric surgery has become a research hotspot. At the same time, other studies have shown that taking probiotics or digestive enzymes may improve gastrointestinal symptoms and improve quality of life after bariatric surgery. Therefore, the purpose of this study was to determine the ability of probiotics to prevent gallstone formation after bariatric surgery and to evaluate the impact of oral probiotics on quality of life in patients after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving bariatric surgery for morbid obesity
* Patiets at ages between 20 to 60 y/o
* Patients willing to follow up regulary after bariatric surgery

Exclusion Criteria:

* Patients having gallstones before bariatric surgery
* Patients refusing taking probiotics or refusing regular follow up after bariatric surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of gallstones in bariatric surgery patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Linglong Yingcheng Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No